CLINICAL TRIAL: NCT07150741
Title: The Effect of Exercise-Assisted Ergonomic Training on Pain, Sleep Quality, and Anxiety Levels in Nursing Students: A Randomized Controlled Trial
Brief Title: Exercise-Assisted Ergonomic Training for Pain, Sleep, and Anxiety in Nursing Students: RCT
Acronym: EASE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Necibe Dağcan, Assistant Professor of Nursing, Kutahya Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KutahyaHSU-NECİBE-DAĞCAN-0007
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pain; Sleep; Anxiety State
Keywords: Pain, Sleep Quality, Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups. The intervention group will receive exercise-assisted ergonomic training, including theoretical lectures and practical exercise sessions, while the control group will continue with the standard nursing curriculum without additional ergonomic or exercise support. Each participant will remain in their assigned group throughout the study, and outcomes will be compared between the two groups.
Who Masked: Outcomes Assessor
Masking Description: Participants and care providers are aware of group assignments. Data collection and outcome assessment will be conducted by a second researcher who is blinded to group allocation. The third researcher performing statistical analyses will also be blinded to group identity to minimize bias in outcome evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive exercise-assisted ergonomic training over 4 weeks. The program includes two theoretical training sessions covering ergonomics, posture analysis, body mechanics, ergonomic risks in nursing, and recommended exercises. In addition, participants will complete eight practical exercise sessions via videos (2 per week, 30-40 minutes each) including warm-up, stretching, strengthening, balance, and posture exercises. The intervention is supervised by an exercise expert to ensure proper technique and safety.
  Interventions: Behavioral: Exercise-Assisted Ergonomic Training
- Control group (No Intervention): Participants will continue with their standard nursing curriculum and will not receive additional ergonomic or exercise training during the study period.

INTERVENTIONS:
Behavioral: Exercise-Assisted Ergonomic Training — The program includes structured ergonomic and exercise activities designed to improve posture, reduce musculoskeletal pain, enhance sleep quality, and decrease anxiety levels among nursing students. Theoretical lectures cover ergonomics principles, postural assessment, body mechanics, and ergonomic risks in nursing. Practical sessions are delivered via video twice a week for 4 weeks, each lasting 30-40 minutes, including warm-up, stretching, strengthening, balance, and posture exercises. The intervention is supervised by an exercise specialist to ensure safety and proper technique.
  Other Names: Ergonomic Training + Exercise Program
  Arms: Intervention Group

SUMMARY:
This randomized controlled trial aims to evaluate the effect of exercise-assisted ergonomic training on pain, sleep quality, and anxiety levels among nursing students. The study population consists of students enrolled in the Nursing Department of Kütahya Health Sciences University. Sixty participants will be recruited according to inclusion criteria and randomly assigned into intervention and control groups.

The intervention group will receive a structured ergonomic training program combined with exercise sessions, including theoretical lectures and practical exercise videos delivered twice a week for four weeks. The control group will continue with their standard nursing curriculum without additional ergonomic or exercise support. Data will be collected using the Numeric Pain Rating Scale, Pittsburgh Sleep Quality Index, and State Anxiety Inventory before and after the intervention.

The study is expected to provide evidence on the effectiveness of ergonomic and exercise-based strategies in reducing pain, improving sleep quality, and lowering anxiety among nursing students, supporting the integration of such programs into nursing education.

DETAILED DESCRIPTION:
Objective:

This study aims to evaluate the effect of exercise-assisted ergonomic training on pain, sleep quality, and anxiety levels among nursing students.

Study Design:

This is a randomized controlled experimental trial. Sixty nursing students who meet inclusion criteria and volunteer to participate will be randomly assigned to either the intervention group (Group A) or control group (Group B), with 30 participants per group. Randomization will be performed using computer-assisted software (www.randomization.com

).

Intervention:

Theoretical Training: The intervention group will receive two theoretical training sessions covering ergonomics, posture analysis, body mechanics, ergonomic risks in nursing, and recommended exercises.

Practical Exercise Sessions: Over four weeks, participants will complete eight exercise sessions (2 per week, 30-40 minutes each) via videos demonstrating warm-up, stretching, strengthening, balance, and posture exercises. The sessions will be supervised by an exercise expert to ensure safety and proper technique.

The control group will continue with the standard nursing curriculum without additional ergonomic or exercise support.

Data Collection:

Data will be collected before and after the intervention using:

Demographic Characteristics Form

Numeric Pain Rating Scale

Pittsburgh Sleep Quality Index

State Anxiety Inventory

Blinding and Bias Prevention:

Participants will be blinded to the group assignments. Data collection will be conducted by a second researcher unaware of the group allocations, and a third researcher will analyze the data while blinded to group identity. CONSORT guidelines will be followed in reporting the results.

Expected Outcomes:

The study is expected to provide evidence on the effectiveness of exercise-assisted ergonomic training in reducing pain, improving sleep quality, and lowering anxiety levels among nursing students, supporting the integration of ergonomic and exercise-based strategies in nursing education.

ELIGIBILITY:
Inclusion Criteria:

* Being a student in the Nursing Department of Kütahya Health Sciences University.
* Willingness to participate in the study voluntarily.
* No chronic diseases preventing exercise (e.g., COPD, heart failure).
* No hearing impairments.
* No psychiatric diagnosis (e.g., major depression, anxiety disorders) and not using related medications.
* Ability to use a smartphone (iOS or Android) and have internet access.
* No neurological, systemic, or psychiatric disorders.

Exclusion Criteria:

* Students unwilling to participate in the study.
* Developing any health problem during the intervention period.
* Unable to continue participation for any reason.
* Voluntarily withdrawing from the study.
* Pain level above 5 on the Numeric Pain Rating Scale at baseline; such participants will be referred to a physiotherapist.
* Any adverse events during exercise sessions (e.g., sudden pain, dizziness, fatigue, blood pressure changes) will result in immediate cessation of the exercise, monitoring of the participant, and referral to the nearest healthcare facility if necessary. Emergency first aid will be provided if needed, and the responsible researcher will contact the relevant health services immediately.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Baseline and 4 weeks after intervention completion
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS) before and after the 4-week exercise-assisted ergonomic training program.

SECONDARY OUTCOMES:
Sleep Quality | Baseline and 4 weeks after intervention completion
  Sleep quality will be measured using the Pittsburgh Sleep Quality Index (PSQI) at baseline and after 4 weeks of intervention.
Anxiety Level | Baseline and 4 weeks after intervention completion
  State anxiety will be measured using the State Anxiety Inventory (SAI) at baseline and after 4 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Necibe DAĞCAN ŞAHİN, PhD, Principal Investigator — Kütahya Health Sciences University, Faculty of Health Sciences; Yiğit ŞAHİN, MSc, Study Director — Kütahya Dumlupınar University, Faculty of Sport Sciences; Mustafa Said ERZEYBEK, Assoc. Prof., Study Director — Kütahya Dumlupınar University, Faculty of Sport Sciences
Locations (1):
- Necibe, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Not applicable. Individual participant data will not be shared.